CLINICAL TRIAL: NCT06669481
Title: Semiquantitative 131I-MIBG Scintigraphy Predicts Intraoperative Blood Pressure Fluctuation in Patients Undergoing Surgery for Pheochromocytoma and Paraganglioma
Brief Title: Correlation Between Preoperative Images of PPGL and Intraoperative Hemodynamics
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: K5426; National High Level Hospital C (Other Grant/Funding Number: 2022-PUMCH-B-071)
Record Dates: First submitted 2024-10-30; First posted 2024-11-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2023-04

CONDITIONS: Pheochromocytoma; Paraganglioma
MeSH Terms: conditions — Pheochromocytoma; Paraganglioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Semiquantitative 131I-MIBG Scintigraphy Assessment — Patients received thyroid blockade using solution of potassium iodide before the examination. After intravenous administration of 111 MBq of 131I-MIBG, whole body planar images were acquired at 24 hours (Day 1) and 48 hours (Day 2), respectively.

SUMMARY:
This is a retrospective observational cohort study involving patients with suspected PPGLs who underwent 131I-MIBG scanning and surgical treatment between January 2020 and April 2023. The objective is to evaluate the correlation between MIBG imaging score and intraoperative hemodynamic fluctuations.

DETAILED DESCRIPTION:
This is a retrospective observational cohort study involving patients with suspected PPGLs who underwent 131I-MIBG scanning and surgical treatment between January 2020 and April 2023. The objective is to evaluate the correlation between MIBG imaging score and intraoperative hemodynamic fluctuations.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected PPGLs who received 131I-MIBG scintigraphy and were treated by surgery

Exclusion Criteria:

* 1) surgery was performed more than 6 months after 131I-MIBG scintigraphy; 2) tumor located in bladder where radioactive urine would influence assessment of tumor; 3) tumor was not resected as a whole; 4) resected tumor was not PPGLs confirmed by pathology; 5) 131I-MIBG scintigraphy images or intraoperative BP was not available for assessment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with suspected PPGLs who received 131I-MIBG scintigraphy and were treated by surgery
Sampling Method: Non-Probability Sample
Enrollment: 159 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Difference of SBP ARV and MAP ARV in Different Groups | Intraoperative systolic blood pressure (SBP) and diastolic blood pressure (DBP) were recorded automatically in a 5 min interval from the beginning to the end of surgery.
  Mean arterial pressure (MAP) was calculated with the formula: MAP=1/3*SBP+2/3*DBP. ARV, which was defined as the average of absolute difference between successive BP values

CONTACTS AND LOCATIONS:
Locations (1):
- Peking union medical college hospital, Beijing, Beijing Municipality, China